CLINICAL TRIAL: NCT00439829
Title: Synchronization of Follicle Wave Emergence and Ovarian Stimulation in Women With a History of Poor Ovarian Response to Treatment
Brief Title: Synchronization of Follicle Wave Emergence and Ovarian Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Angela Baerwald - Scientific Investigator, Reproductive Biology Research Unit, Dept OB/GYN, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-REB 06-03; HlthCanadaFile#9427-U0208-47C
Record Dates: First submitted 2007-02-13; First posted 2007-02-26 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Infertility
Keywords: follicle; ovary; poor responder; stimulation; follicle wave emergence
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Luteinizing Hormone, beta Subunit; cetrorelix

ARMS (2):
- 1 (Experimental): Initiation of ovarian stimulation therapy on day 1 (i.e., first day of menses)
  Interventions: Drug: Gonal F; Drug: Luveris; Drug: Cetrotide; Drug: hCG
- 2 (Active Comparator): Initiation of ovarian stimulation therapy on day 4 (day 1= first day of menses)
  Interventions: Drug: Gonal F; Drug: Luveris; Drug: Cetrotide; Drug: hCG

INTERVENTIONS:
Drug: Gonal F — * 450 IU Gonal-f (Serono Canada) subcutaneously daily (225 IU BID; injections to be given after bloodwork).
  * Dosing to begin on day 1 or day 4 (day 1=first day of menses), continuing until administration of human Chorionic Gonadotropin (hCG; see below).
  * Gonal-f dose may be further reduced, at the discretion of the study physician, to minimize the risk of OHSS.
Drug: Luveris — * 0.250 mg Cetrotide (Serono Canada) and 75 IU Luveris (Serono Canada) subcutaneously daily when one or more of the following conditions are met:
    * leading follicle is > 13 mm in diameter
    * if 6 or more follicles develop to > 10 mm and E2 > 1000 pmol/L
  * Dosing to continue until administration of hCG (see below).
Drug: Cetrotide — * 0.250 mg Cetrotide (Serono Canada) and 75 IU Luveris (Serono Canada) subcutaneously daily when one or more of the following conditions are met:
    * leading follicle is > 13 mm in diameter
    * if 6 or more follicles develop to > 10 mm and E2 > 1000 pmol/L
  * Dosing to continue until administration of hCG (see below).
Drug: hCG — - 10,000 IU hCG (Pharmaceutical Partners of Canada Inc.) subcutaneously when:
  o > 3 follicles are > 17 mm in diameter

SUMMARY:
The objective of the study is to elucidate the effect of synchronizing initiation of ovarian stimulation treatment with follicular wave emergence in poor responder patients undergoing IVF/ICSI and ET. We hypothesize that initiating treatment on day 1 versus day 4 of the cycle will increase the number of follicles recruited and oocytes retrieved.

DETAILED DESCRIPTION:
Sample Population Eligible patients undergoing IVF or ICSI for the treatment of infertility in the Assisted Reproductive Technologies Center at the University of Saskatchewan (ARTUS; Department of Obstetrics, Gynecology and Reproductive Sciences) in Saskatoon, Saskatchewan and the Genesis Fertility Centre in Vancouver, British Columbia will be identified by study physicians and nurses. Patients with a history of poor response to ovarian stimulation therapy in a previous IVF or ICSI cycle, who have already decided to undergo a subsequent treatment cycle, will be contacted by a study physician and offered enrolment into the study. Patients exhibiting all inclusion criteria and no exclusion criteria will be eligible to participate.

Inclusion Criteria:

* Informed consent obtained
* Age of 43 years or younger
* 18<BMI<35
* History of poor response to ovarian stimulation as determined by:
* previously cancelled oocyte retrieval procedure due to < 4 follicles greater than 12 mm on ultrasound OR
* < 3 mature oocytes
* Physical exam performed within the past 12 months
* Normal or corrected levels of TSH and Prolactin within the past 12 months
* Has not taken ovarian suppression therapy within 1 month of initiating study drug

Exclusion Criteria:

* Chronic medical conditions such as renal failure
* Documented ovarian failure
* Presence of only one ovary
* Serum Day 3 FSH > 12 IU/L within the past 6 months
* Ovaries inaccessible transvaginally
* Concomitant glucocorticoid use
* Ongoing pregnancy
* Any contraindications to ovarian stimulation treatment
* Participation in an investigational drug trial in the 30 days prior to the pre-study visit

Cycle Cancellation Criteria:

* The development of < 3 follicles > 12 mm.

Sample Size A sample size of 80 women (40 women per treatment group) has been chosen. This calculation was based on a standard deviation of 3.0 in each treatment group, a significance level of 0.05 (2-tailed test), a mean difference of 2.0 follicles and a power of 80%. The standard deviation used in the power calculation was based on similar studies performed in domestic animal species. Approximately 120 IVF/ICSI cycles are performed each year in the Department of Obstetrics, Gynecology and Reproductive Sciences at the University of Saskatchewan and approximately 600 cycles are performed at the Genesis Fertility Centre. Approximately 5-10% of patients are proven poor responders. Thus, with an anticipated 75% recruitment rate, we expect to recruit 80 patients in the study over a 24 month period. It is expected that 25% of research subjects will be enrolled at the ARTUS Centre and 75% of subjects will be enrolled at the Genesis Fertility Centre.

Study Procedures Women who are believed to be eligible for the study will be asked to visit the Assisted Reproductive Technologies Center at the University of Saskatchewan (ARTUS) or the Genesis Fertility Centre in Vancouver, British Columbia for a pre-study appointment. At this visit, inclusion and exclusion criteria will be reviewed. If patients meet all study criteria, consent will be obtained and each woman will be randomized to either the control group (i.e. treatment starting on day 4) or experimental group (i.e., treatment starting on day 1). A medical history and vital signs will be performed. Study drug administration, diary card use and potential adverse reactions will be reviewed at the pre-study visit. Diary cards will be used to monitor study drug administration, adverse reactions, and concomitant medications used during the study. Diary cards will be reviewed with the patient by study personnel throughout the duration of the study. Serious adverse events will be reported by the investigators to the drug safety group of the study drug manufacturers and the Biomedical Research Ethics Board, in accordance with Tri-Council Policy guidelines.

All patients will be instructed to call the clinic on day 1 of menses. If menses begins before 6 pm, that day will be considered day 1. If menses begins after 6 pm, the next day will be considered day 1. Women randomized to the day 1 treatment group will be instructed to begin ovarian stimulation therapy (Gonal-f, Serono Canada) on day 1 and visit the clinic to undergo their first transvaginal ultrasound examination on day 2. Women randomized to the day 4 treatment group will be instructed to begin ovarian stimulation on day 4 and visit the clinic on day 4 for their first transvaginal ultrasound examination. Ultrasound examinations will be performed to determine the number of follicles developing in the ovaries. Ultrasound examinations will continue every 2-4 days for each woman, as per the normal standard of care. Blood will be drawn intermittently during stimulation to determine serum concentrations of estradiol-17B. Each participant will be asked to perform a home urine pregnancy test before taking their first dose of study medication. If a woman is found to be pregnant, she will be withdrawn from the study.

When a follicle > 13 mm is detected OR if 6 or more follicles > 10 mm develop and E2 is > 1000 pmol/L, women will be instructed to begin taking a Gonadotropin Releasing Hormone Antagonist (Cetrotide, Serono Canada) and recombinant Luteinizing Hormone (Luveris, Serono Canada). Gonal F, Cetrotide and Luveris administration will continue daily until human Chorionic Gonadotropin (hCG, Pharmaceutical Partners of Canada Inc.) is administered when > 3 follicles reach > 17 mm in diameter. It is anticipated that the duration of ovarian stimulation therapy will be 8-16 days. Shorter or longer stimulation intervals may result in cycle cancellation. Oocytes will be isolated, evaluated and fertilized following hCG administration, according to the normal standard of care.

The type and dose of stimulation therapy will be standardized among women as noted in Appendix B. Women will be asked to visit the clinic for a follow-up appointment with the physician and study nurse approximately 4 weeks after the oocyte retrieval. Adverse events, concomitant medications and diaries will be reviewed at this time. After the follow-up appointment, women will have completed all study-related procedures. Adverse events persisting at the time of study completion will be followed as deemed medically appropriate.

All procedures performed in this study adhere to Good Clinical Practice guidelines. The only procedures that differ from those carried out for routine patient care are the initiation of ovarian stimulation therapy on day 1, the urine pregnancy test prior to initiating therapy and the completion of diary cards by the patients to monitor study drug administration, adverse events and concomitant medications.

Study Endpoints

Primary study endpoints include:

* number of follicles > 15 mm on day of hCG
* peak serum estradiol concentrations

Secondary study endpoints include:

* number of antral follicles (day 1 or day 4)
* number of follicles aspirated
* number of oocytes obtained
* oocyte morphology
* fertilization rates
* number of viable embryos (day 3 and day 5)
* blastocyst rate
* number of embryos transferred
* clinical pregnancy rate (serum ß-hCG)

All study endpoints will be compared between women in the control versus experimental group. An interim analysis will be performed by the study investigators once 40 patients have completed study procedures. The overall incidence of Ovarian Hyperstimulation Syndrome (OHSS) requiring hospitalization in women undergoing IVF/ICSI is approximately 3%. Therefore, in 40 normal responder patients we would expect an incidence of OHSS-related hospitalization to be approximately 1.2%. If more than 1 patient in each treatment group has been admitted to the hospital for OHSS after 40 women have completed study procedures, the study will be reviewed for possible termination.

Foreseeable Risks and Discomfort

Potential risks during study participation include:

* discomfort during transvaginal ultrasound examination
* discomfort and bruising at the site of venipuncture
* redness, swelling and discomfort at the drug injection site
* ovarian hyperstimulation

In 1-10% of normally-responding patients, ovarian hyperstimulation syndrome (OHSS) occurs in which too many follicles develop, placing the woman at risk for hospitalization. Because a suboptimal number of follicles develop in women who respond poorly to ovarian stimulation therapy, we believe that the risk of ovarian hyperstimulation is extremely low to zero. However, because we cannot predict the outcome of initiating therapy on day 1 of the menstrual cycle, we cannot guarantee that hyperstimulation will not occur.

All of the above-mentioned risks are related to current standard of care for IVF. The risks of OHSS will be minimized by adherence to the usual standard of care for ovarian stimulation monitoring. Patients felt to be at risk for developing OHSS will have their dose of exogenous FSH and hCG therapy dropped, as per the usual standard of care.

In the event that patients become ill or injured as a result of participating in this study, necessary medical treatment will be made available at no additional cost to the patient. By signing the consent form, patients do not waive any of their legal rights.

Benefits There are no guaranteed benefits for women participating in this study. However, if our hypothesis is proven, women may benefit from an increased number of recruited follicles. We anticipate that the results of this study will increase our understanding of poor response to ovarian stimulation, and lead to the development of better treatments for couples undergoing IVF/ICSI and ET in the future.

Costs Partial drug coverage will be provided by Serono Canada Inc. to participants in this study.

Confidentiality All participants will be identified in the study by their initials and assigned patient study number. Only study personnel will have access to study-related records during the conduct of the study. The contents of study related records will not be available to any party other than the University of Saskatchewan Ethics Board, the study sponsor, and government regulatory agencies unless required by law. A report of the results of this study may be made to Health Canada (HC) and the Food and Drug Administration (FDA, USA) while maintaining confidentiality of patient identification. The results of this study may also be used for medical and scientific publications but patient identity will not be disclosed. Study files will be archived by the scientific investigator for 25 years at Royal University Hospital.

Voluntary Participation/Withdrawal from Study Participation in this study is voluntary. Patients may decide not to participate or may withdraw at any time. Refusal to participate in, or withdrawal from, the study will not affect the future medical care of the patient.

Participation in this study may be ended at any time, without patient consent. Reasons may include, but are not limited to, patient's failure to follow study instructions, the appearance of side effects, or study cancellation due to administrative reasons. If < 3 follicles develop to a diameter of 12 mm or larger, the patient will be withdrawn from the study and the IVF/ICSI cycle may be cancelled.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Age of 43 years or younger
* 18 < BMI < 35
* History of poor response to ovarian stimulation as determined by:

  * previously cancelled oocyte retrieval procedure due to < 4 follicles greater than 12 mm on ultrasound OR
  * < 3 mature oocytes
* Physical exam performed within the past 12 months
* Normal or corrected levels of TSH and Prolactin within the past 12 months
* Has not taken ovarian suppression therapy within 1 month of initiating study drug

Exclusion Criteria:

* Chronic medical conditions such as renal failure
* Documented ovarian failure
* Presence of only one ovary
* Serum Day 3 FSH > 12 IU/L within the past 6 months
* Ovaries inaccessible transvaginally
* Concomitant glucocorticoid use
* Ongoing pregnancy
* Any contraindications to ovarian stimulation treatment
* Participation in an investigational drug trial in the 30 days prior to the pre-study visit

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
number of follicles greater than or equal to 15 mm on day of hCG | March 2009
peak serum estradiol concentrations | March 2009

SECONDARY OUTCOMES:
number of antral follicles (day 1 or day 4) | March 2009
number of follicles aspirated | March 2009
number of oocytes obtained | March 2009
oocyte morphology | March 2009
fertilization rates | March 2009
number of viable embryos (day 3 and day 5) | March 2009
blastocyst rate | March 2009
number of embryos transferred | March 2009
clinical pregnancy rate (serum ß-hCG) | March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Baerwald, PhD, Study Director — Dept OB/GYN, University of Saskatchewan; Allison M Case, MD FRCSC, Principal Investigator — Dept OB/GYN, University of Saskatchewan
Locations (2):
- Canada (2):
  - Genesis Fertility Centre, Vancouver, British Columbia
  - Department of Obstetrics, Gynecology and Reproductive Sciences, University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128
- [Derived] Baerwald A, Anderson P, Yuzpe A, Case A, Fluker M. Synchronization of ovarian stimulation with follicle wave emergence in patients undergoing in vitro fertilization with a prior suboptimal response: a randomized, controlled trial. Fertil Steril. 2012 Oct;98(4):881-7.e1-2. doi: 10.1016/j.fertnstert.2012.06.051. Epub 2012 Jul 20. PMID 22819187